CLINICAL TRIAL: NCT07210645
Title: Development of a Power Training Program to Improve Mobility in Older Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRD8-001-24W; 25-1070 (Other: COMIRB)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Physical Deconditioning; Mobility Decline
Keywords: power training; mobility; older adult; user-centered design

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 2 groups: Group 1 (Gerofit power training) will receive the intervention for 6 months, and Group 2 (Gerofit standard of care) will receive standard of care for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gerofit Power Training Intervention (Experimental): This group will be randomized to receive Gerofit power training intervention for 6 months. They will receive power training as part of each Gerofit exercise session. Gerofit exercise sessions also include aerobic, flexibility, and balance training.
  Interventions: Other: Gerofit Power Training
- Gerofit Standard of Care (Active Comparator): This group will be randomized to receive standard of care exercise Gerofit exercise prescription for 6 months. Standard of care exercise for the Gerofit program includes combined aerobic, strength, flexibility and balance training.
  Interventions: Other: Gerofit Standard of Care

INTERVENTIONS:
Other: Gerofit Power Training — Gerofit Power Training will include a power training exercise prescription which will focus on having participants perform concentric portions of each resistance exercise as fast and as safely as possible with the eccentric component performed in a slow and controlled manner. The target dose of the power training intervention is 40-60% of the participant's 1-repetition maximum for 4-6 repetitions across 3-6 sets for each exercise. Exercises will focus on the major groups of the upper and lower body. All other Gerofit program components (balance, aerobic, and flexibility) will be consistent with the standard of care group. Sessions will be the same duration as the standard of care Gerofit group (60-75 minutes). The power training and standard of care groups will only differ in the form of resistance training performed.
  Arms: Gerofit Power Training Intervention
Other: Gerofit Standard of Care — Gerofit standard of care is a 60-75 minute multimodal exercise program which includes 20-30 minutes of aerobic training, traditional strength training of the major upper and lower body muscle groups (1-3 sets of 8-12 repetitions at moderate load), flexibility training and balance training.
  Arms: Gerofit Standard of Care

SUMMARY:
The overall purpose of this study is to develop a power training intervention in partnership with Veterans participating in Gerofit and to evaluate the program's acceptability, feasibility, and preliminary participant outcomes (leg power, physical function and self-report participation).

DETAILED DESCRIPTION:
The overall purpose of this project is to co-design a power training intervention for Veterans engaged in Gerofit and to assess its feasibility, acceptability, and preliminary participant outcomes. Gerofit Veterans and exercise providers will participate in co-designing the power training intervention through interviews and feedback sessions. The power training program developed will be tested in the subsequent randomized feasibility pilot. This pilot aims to evaluate the feasibility, acceptability, and preliminary outcomes of a power training program in older Veterans participating in Gerofit using an explanatory sequential mixed methods design. Veterans newly enrolled in the Gerofit program will be randomized into power training and standard of care groups and will participate in exercise sessions over 6 months. Feasibility and acceptability will be assessed by Veteran adherence to program components and by validated surveys. Quantitative data collection will inform qualitative interviews with Veterans on the acceptability and feasibility of the power training program at its completion. Clinical outcomes will be collected (leg power, physical function, and self-report participation) at baseline, 3 months and 6 months and will be compared between the Gerofit power training and Gerofit standard of care groups. Study findings will lead to the development of a power training program that optimally meets Veteran and Gerofit program needs. In addition, study outcomes will guide implementation of a power training program into Gerofit programs aimed at enhancing mobility outcomes in older Veterans.

ELIGIBILITY:
Inclusion Criteria:

Pilot Study Criteria:

* Veterans 65 years of age and older
* New enrollees of the Rocky Mountain Regional Gerofit Program
* ability to function independently in a group setting

Exclusion Criteria:

* inability to perform basic activities of daily living
* oxygen dependency
* unstable cardiac disease
* moderate to severe cognitive impairment (Montreal cognitive assessment scores < 24)
* proliferative diabetic retinopathy
* relative exclusions for participation in the in-person Gerofit exercise program including: open wounds, incontinence, and lack of transportation
* inability to ambulate
* progressive neurological diagnoses (e.g. Amyotrophic lateral sclerosis, Parkinson's disease, multiple sclerosis)
* individuals with planned orthopedic surgeries in the next 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-06 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | assessed at 3-months (primary endpoint) and 6 months in both intervention and standard of care groups
  Adherence will be measured as a proportion of the number of sessions attended out of the number prescribed per protocol.

SECONDARY OUTCOMES:
Retention | assessed at 3-months (primary) and 6 months
  Retention will be tracked as part of feasibility and to inform a future trial. Retention will be measured as the proportion of Veterans who complete all outcome measure timepoints out of the total who complete baseline measures.
Feasibility | assessed at 3-months (primary) and 6 months
  Feasibility will be measured through a validated survey: Feasibility of Intervention Measure which consists of 4 items rated on a 5-point Likert scale ranging from (1) completely disagree to (5) complete agree. Higher scores indicate greater feasibility of the program. Measure will only be collected in the intervention group.
Acceptability | assessed at 3-months (primary) and 6 months
  Acceptability will be measured through a validated survey: Theoretical Framework of Acceptability Measure which consists of 8 items rated on a 5-point Likert scale ranging from (1) did not like, high burden to (5) strongly liked, low burden. Higher scores indicate greater acceptability of the program. Measure will only be collected in the intervention group.
Leg Press Power | baseline, 3-months and 6 months
  Leg power will be evaluated using previously validated methods in older adults at 40% and 70% of the Veterans 1-repetition maximum over 5 repetitions. Scores are continuous, higher scores indicate greater leg power (better outcome).
4 stair climb power test (4SCPT) | baseline, 3-months and 6 months
  Power in Watts will be measured using a valid and reliable test which calculates power from time, body weight and stair height when participants climb 4 steps as fast as possible. Scores are continuous, higher scores indicate greater leg power (better outcome).
Gait speed | baseline, 3-months and 6 months
  This is a functional test of mobility. Participants will be timed while walking at self-selected and fast speeds for 10 meters. Gait speed in meters per second will calculated for self-selected and fast gait speeds. Scores are continuous, higher scores indicate greater greater gait speed and mobility (better outcome).
Late Life Function and Disability Instrument (LLFDI) | baseline, 3-months and 6 months
  Participants will complete this valid and reliable self-report measure of physical function (32 items) and disability (16 items). Raw summary scores are transferred to scaled summary scores on a 0-100 scale with higher scores indicated greater function and greater participation in life tasks.
30 second chair rise | baseline, 3-months and 6 months
  This is a functional test of leg strength and power. Participants are asked to stand up and sit down as many times as they can in 30 seconds from a standard height chair. Scores are continuous, higher scores indicate greater leg strength and power (better outcome).
arm curl test | baseline, 3-months and 6 months
  This is a functional performance test for upper body strength and is performed on each arm (one arm at a time). It requires the participant to perform as many arm curls (bicep curls) as possible in 30 seconds. Males use an 8lb weight and females use a 5 lb weight. Scores are continuous, and higher scores indicate greater arm strength (better outcome).
6 minute walk test | baseline, 3-months and 6 months
  This is a functional test of aerobic capacity. Participants walk as far as they can along a preset track in 6 minutes. Score is the maximal distance walked in 6 minutes, measured in meters. Scores are continuous, and higher scores indicate greater aerobic capacity (better outcome).
Leg press strength | baseline, 3-months and 6 months
  This is a test of lower body muscle strength. Participants will perform a 1-repetition maximum leg press test where they press the heaviest load they can 1 time through their full range of motion with good form. The test is scored in pounds. Scores are continuous, and higher scores indicate greater leg strength (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Mattie E Pontiff, PT, DPT, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No